CLINICAL TRIAL: NCT04053673
Title: A Phase 1, First-in-human Study of the Safety, Single- and Multiple-Dose Pharmacokinetics, and Preliminary Activity of Escalating Doses of RBN-2397, an Oral PARP7 Inhibitor, in Patients With Solid Tumors
Brief Title: Phase 1 Study of RBN-2397, an Oral PARP7 Inhibitor, in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ribon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RBN-2397-19-001
Record Dates: First submitted 2019-08-05; First posted 2019-08-12 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumor, Adult
Keywords: Phase 1; PARP7 inhibition; First in Human; Solid Tumors; Interferon

STUDY DESIGN:
Intervention Model Description: Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RBN-2397 (Experimental): Dose Escalation: Multiple doses of RBN-2397 for oral administration Dose Expansion: Oral dose of RBN-2397 as determined during Dose Escalation
  Interventions: Drug: RBN-2397

INTERVENTIONS:
Drug: RBN-2397 — an oral PARP7 Inhibitor

SUMMARY:
RBN-2397 inhibits PARP7, an enzyme that is switched on by cancer stresses, such as the toxins in cigarette smoke. Cancer cells use PARP7 to hide from the immune system by stopping the cell from sending a signal (Type 1 interferon) that tells the immune system that something is wrong and to kill the cell. RBN-2397 has been shown in animal studies to inhibit tumor growth and also shuts down the "don't kill me" signal the tumor is sending to evade the immune system. As a PARP7 inhibitor RBN-2397 is different from drugs inhibiting PARP1, PARP2 and PARP3 enzymes which are approved for the treatment of certain ovarian and breast cancers.

The primary purpose of this study is to determine the maximum tolerated dose (MTD) of orally administered RBN-2397 in patients with advanced or metastatic solid tumors. This study will also evaluate the safety and tolerability of RBN-2397, examine the pharmacokinetics (PK) (measure how the body absorbs, breaks down and eliminates RBN-2397) and investigate whether it has antitumor activity in solid tumor cancers.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, multi-center, open-label, dose-escalation study to:

* Evaluate the safety profile and MTD of RBN-2397 administered orally and establish the RBN-2397 dose(s) and schedule(s) recommended for further investigation in Phase 2
* Characterize the PK profile of RBN-2397
* Identify preliminary antitumor activity.
* Biomarkers and their correlation with response to RBN-2397 and other outcomes will be examined.

Cohorts will follow a traditional 3 + 3 design. After enrollment of the first participant within a cohort, there must be a wait period of at least 1 week before enrollment of additional participants in that cohort. This dose escalation phase of the study is complete.

The study is currently in the Relative Bioavailability and Expansion Cohort(s) phase where approximately 20 participants each will be enrolled to further examine the safety, PK, pharmacodynamics, and antitumor activity of RBN-2397 at the recommended phase 2 dose.

Relative Bioavailability Assessment:

An evaluation of relative bioavailability of a micronized RBN-2397 tablet versus the standard RBN-2397 tablet (manufactured with unmicronized RBN-2397 and used in the dose escalation phase of the study) will be performed as part of the dose escalation phase. Micronized tablets will be used in the Dose Expansion Phase of the study after the relative bioavailability assessment has been completed.

Dose Expansion Phase The recommended phase 2 dose will be investigated in the following cancer types: squamous cell carcinoma of the lung (SCCL), head and neck squamous cell carcinoma (HNSCC), hormone receptor positive (HR+) breast cancer, and PARP7 amplified cancer.

Duration of treatment:

It is anticipated that the minimum study involvement will be one cycle. Participants are eligible to have an indefinite number of additional cycles of treatment if their disease does not progress and they do not have unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation Phase only: Metastatic or advanced-stage solid malignant tumor (which may include "solid" lymphoma [e.g., mantle cell]) for whom no therapy exists that would be curative or might provide clinical benefit.

Dose Expansion Phase Only: Patients with locally advanced or metastatic solid tumors, with at least one measurable lesion as determined by RECIST version 1.1, who have received standard therapy or are intolerant of standard therapy, have progressed following their last prior therapy, and have one of the following tumor types:

* SCCL: Histologically confirmed NSCLC of predominantly squamous cell histology and must have received no more than 3 lines of prior systemic therapy including chemotherapy regimens and/or immune checkpoint inhibitor therapy (combination allowed).
* HNSCC: Histologically confirmed squamous cell carcinoma of the head and neck (either HPV-positive or -negative) and must have received no more than 3 lines of prior systemic immunotherapy and/or chemotherapeutic treatments in the metastatic setting. Includes primary tumor location of the oral cavity, oropharynx, hypopharynx, larynx, and paranasal sinuses (nasopharyngeal carcinoma, skin squamous cell carcinoma, and salivary gland carcinomas are not eligible).
* HR+ breast cancer: Histologically confirmed diagnosis of estrogen receptor (ER) and/or progesterone receptor (PR) positive, HER2-negative adenocarcinoma of breast (as per local laboratory testing) whose disease has failed standard systemic therapy for locally advanced or metastatic disease and must have received no more than 1 prior chemotherapeutic for advanced/metastatic disease.
* PARP7 amplified: Tumor with documented PARP7 (or TIPARP) gene copy amplification as determined by a CLIA certified laboratory test (e.g., FoundationOne CDx) that has failed standard systemic therapy for locally advanced or metastatic disease.

Must agree to undergo tumor biopsy Normal organ and bone marrow function Patient and his/her partner agree to use adequate contraception during and for 3 months after the last study drug dose

Exclusion Criteria:

* Unable to swallow oral medications
* Major surgery within 4 weeks of starting study
* Pregnant or breast-feeding.
* Receiving intravenous antibiotics for an active infection
* Known human immunodeficiency virus (HIV) or hepatitis B or C infection.
* History of a different malignancy unless disease-free for at least 5 years
* Some medications are not allowed while on study. Interested participants will need to inform study doctor of all the medications he/she is taking.
* Herbal medicines, and grapefruit, grapefruit juice, pomegranate juice, star fruit or orange marmalade (made with Seville oranges) are not allowed to be taken during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) | through first treatment cycle (an average of 21 days)
  Incidence of Dose limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
Safety and tolerability | through study completion (an average of one year)
  Grade and frequency of adverse events and serious adverse events
Area under the plasma concentration for tablet manufactured with micronized RBN-2397 relative to unmicronized RBN-2397 (standard tablet) (Relative Bioavailability Cohorts only) | Through Study Day 22
  Area-under-the-curve (AUC inf)
Peak plasma concentration for tablet manufactured with micronized RBN-2397 relative to unmicronized RBN-2397 (standard tablet) (Relative Bioavailability Cohorts only) | Through Study Day 22
  Cmax
Antitumor activity that may be associated with RBN-2397 treatment assessed by CT/MRI Response Evaluation Criteria for Solid Tumors (RECIST) Criteria v1.1 | Every 6-8 weeks; through study completion (an average of one year)
  Objective response rate (ORR)
Antitumor activity that may be associated with RBN-2397 treatment | Every 6-8 weeks; through study completion (an average of one year)
  Disease control rate (DCR)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Johnson, MD, Principal Investigator — Tennessee Oncology
Locations (15):
- United States (11):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - SCRI-Denver/HealthOne, Denver, Colorado
  - Yale Cancer Center, Yale University, New Haven, Connecticut
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - SCRI-Sarasota/Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - SCRI-Nashville/Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Spain (4):
  - Hospital Quironsalud Barcelona - NEXT Oncology, Barcelona
  - Vall d'Hebron, Barcelona
  - Hospital Quironsalud Madrid - NEXT Oncology, Madrid
  - Hospital Clinic Universitario Biomedical Research institute INCLIVA, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen MS, Chang P. Insights into the biogenesis, function, and regulation of ADP-ribosylation. Nat Chem Biol. 2018 Feb 14;14(3):236-243. doi: 10.1038/nchembio.2568. PMID 29443986
- [Background] Gozgit JM, Vasbinder MM, Abo RP, Kunii K, Kuplast-Barr KG, Gui B, Lu AZ, Molina JR, Minissale E, Swinger KK, Wigle TJ, Blackwell DJ, Majer CR, Ren Y, Niepel M, Varsamis ZA, Nayak SP, Bamberg E, Mo JR, Church WD, Mady ASA, Song J, Utley L, Rao PE, Mitchison TJ, Kuntz KW, Richon VM, Keilhack H. PARP7 negatively regulates the type I interferon response in cancer cells and its inhibition triggers antitumor immunity. Cancer Cell. 2021 Sep 13;39(9):1214-1226.e10. doi: 10.1016/j.ccell.2021.06.018. Epub 2021 Jul 22. PMID 34375612